CLINICAL TRIAL: NCT05056623
Title: Effectiveness of a Dyadic Pain Management Program for Community-dwelling Older Adults with Chronic Pain: a Cluster Randomized Controlled Trial
Brief Title: Effectiveness of a Dyadic Pain Management Program for Community-dwelling Older Adults with Chronic Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Collaborators: Health and Medical Research Fund (Other Government); Shatin Hospital (Other); The Hong Kong Polytechnic University (Other); The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Mimi TSE Mun Yee, Professor, Hong Kong Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: DPM
Record Dates: First submitted 2021-03-24; First posted 2021-09-24 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Chronic Pain; Elderly; Informal Caregivers; Dyadic Intervention
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dyadic pain management program (Experimental): The DPM is an 8-week group-based program. The DPM included 4 weeks of center-based, face-to-face activities and 4 weeks digital-based activities delivered via a WhatsApp group.
  Interventions: Behavioral: Dyadic pain management program
- Usual care and pain management pamphlet (Other): The participants in the control group will receive the usual care and a pain management pamphlet.
  Interventions: Other: Usual care and pain management pamphlet

INTERVENTIONS:
Behavioral: Dyadic pain management program — Face-to-face part: The DPM will start with 20-30 minutes of physical exercise supervised by research assistant, followed by 20-minutes of pain management education. Communication skills regarding the practice of various pain management techniques by the participants and their caregivers will be taught. At the end of the session, the caregiver and research assistant will help the older adults to make portfolio entries on the activities of the day, to help them recall the various pain-relief methods learned in each class.
  Home-based part: An exercise book will be given to guide them in performing exercises at home. It is recommended to perform 30 minutes of exercise, 3 times a week, at home and the more frequent the exercise time, the better.
  All participants will join a WhatsApp group to receive teaching materials and videos of the physical exercises learned, for practice at home. The team will produce compact disc (CD) with the exercise video clips to the dyads for revision.
  Arms: Dyadic pain management program
Other: Usual care and pain management pamphlet — Usual care and pain management pamphlet
  Arms: Usual care and pain management pamphlet

SUMMARY:
Objective: To evaluate the effectiveness of a dyadic pain management program (DPM) in reducing pain and psychological health symptoms, improving pain self-efficacy, quality of life, and physical function in older adults.

Hypothesis: DPM is more effective in reducing pain and psychological health symptoms, improving pain self-efficacy, quality of life, and physical function among older adults than the usual care, upon completion of the DPM (week 8) and over time (week 16).

Design and subjects: Clustered randomized controlled trial with neighborhood elderly centers (NEC) as cluster; 150 dyads (one older adults and his/her caregiver as one dyad) will be recruited from 22 NEC clusters. Each NEC will be randomly allocated to experimental group (receive DPM), control group (receive usual care and pain management pamphlet).

Study instruments: Brief Pain Inventory; Pain Self-Efficacy Questionnaire; Short Form Health Survey-12; Depression, anxiety & stress; Caregiver Burden Inventory; 6-minute walk test and process evaluation.

Intervention: DPM, each session includes exercise, interactive pain management education, practices on non-drug techniques and using a WhatsApp (WhatsApp Messenger) group to encourage home-based exercise and practice of non-drug methods.

Outcome measures: Pain intensity, pain self-efficacy, perceived health-related quality of life and experience in participating DPM, to be collected at baseline (T0), week 8 (T1), and week 16 (T2).

Data analysis: Multilevel regression and/or Generalized Estimating Equation will be used for within-group and between- group comparisons.

DETAILED DESCRIPTION:
The DPM is an 8-week group-based program. The DPM included 4 weeks of center-based, face-to-face activities and 4 weeks digital-based activities delivered via a WhatsApp group. An 80% participation rate in the face-to-face activities will be regarded as completion of the DPM. Timely make-up sessions will be arranged for those unable to attend the scheduled session.

ELIGIBILITY:
Older adults / Participants: Inclusion criteria

* Aged 60 or above who are mainly cared for by an informal caregiver and willing to participate the DPM together
* scored >6 in the Abbreviated Mental Test; a cut-off point of 6 is valid in differentiating between normal and abnormal cognitive functions for geriatric clients29 Can understand Cantonese
* Have a history of non-cancer pain in the past 6 months
* Have a pain score of at least 2 on the Numeric Rating Scale (0-11 numeric scale)
* Able to take part in light exercise and stretching
* One member of the dyad owns a smart phone and can access the Internet

Older adults / Participants: Exclusion criteria

* Have a serious organic disease or malignant tumor
* Have a mental disorder diagnosed by neurologists or psychiatrists
* Will have further medical/surgical treatment in two months
* Experienced drug addiction18

Informal Caregivers : Inclusion criteria

* Aged 18 or above
* As an informal caregiver for the participating older adult
* scored >6 in the Abbreviated Mental Test; a cut-off point of 6 is valid in differentiating between normal and abnormal cognitive functions for geriatric clients
* Can understand Chinese
* Have a history of non-cancer pain in the past 6 months
* Have a pain score of at least 2 on the Numeric Rating Scale (0-11 numeric scale)
* Able to take part in light exercise and stretching
* Own a smart phone and can assess the internet
* Able to attend the whole sessions in community activity center

Informal Caregivers: Exclusion criteria

* Have serious organic disease or malignant tumor
* Have a history of consciousness or mental disorder diagnosed by neurologists or psychiatrists
* Have a further medical/surgical treatment in two months or have joined in other pain management program
* Experience a drug addiction problem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-07-14 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline pain intensity at week 16 | Baseline to week 16
  The Chinese version of the Brief Pain Inventory will be used to assess the multidimensional nature of pain, including intensity and interference with life activities in the previous 24 hours. Minimum score = 0; Maximum score = 10. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Pain self-efficacy | Baseline (T0), week 8 (T1), week 16 (T2)
  A Chinese version of the Pain Self-Efficacy Questionnaire (PSEQ) will be used to measure self-efficacy in coping with activities despite pain. Minimum score = 0; Maximum score = 60. Higher scores mean a better outcome.
Perceived quality of life | Baseline (T0), week 8 (T1), week 16 (T2)
  The Chinese version of the EuroQoL 5-dimension 5-level version (EQ-5D-5L) will be used to measure quality of life of participants as well as the cost effectiveness of the proposed dyadic pain management program. It is a health-related quality of life measure developed by the EuroQol Group. Minimum score = 0; Maximum score = 100. Higher scores means a better outcome.
Psychological health : Depression, anxiety, & stress | Baseline (T0), week 8 (T1), week 16 (T2)
  The Depression Anxiety Stress Scales 21-items (DASS-21) is a self-administered psychological instrument to evaluate degrees of depression, anxiety, and stress. Minimum score. Minimum score = 0; Maximum score: Depression = 28+, Anxiety = 20+, Stress = 37+. Higher score means a worse outcome.
Physical function: 6-minute walk test | Baseline (T0), week 8 (T1), week 16 (T2)
  A 6-minute walk test to test exercise tolerance in chronic disease.
Caregiver Burden Inventory (for the caregivers only) | Baseline (T0), week 8 (T1), week 16 (T2)
  The Caregiver Burden Inventory comprises 24 items measuring five dimensions of burden related to the caregiving role. Minimum score = 0; Maximum score 96. Higher score means a worse outcome.
Process evaluation | Baseline (T0), week 8 (T1), week 16 (T2)
  A process evaluation will be carried out to identify the strengths and limitations of the intervention from the perspectives of the older adults and their caregivers
Field observations | Each DPM will be observed twice within four sessions when carrying out the DPM through 8-week group-based program
  To monitor the quality of the implementation of the DPM. A total of 48 observations will be conducted by the principal investigator, guided by a fidelity checklist. 9 The checklist indicates the implementation of DPM in terms of four levels: low/not observed; observed to a small degree; observed to a medium degree, and high implementation.
Knowledge and skills acquired in managing pain situations for older adults | Baseline (T0), week 8 (T1), week 16 (T2)
  A questionnaire will be given to the participants in the experimental and control groups regarding their knowledge and skills in managing pain situations. Minimum score = 0, Maximum score = 10. Higher score means a better outcome.
Semi-structured interviews for older adults and their caregivers | Individual interviews will be conducted by the Research Assistant 1 within 2 weeks after T1
  To obtain the widest range of opinions and comments from different perspectives, equal proportions of participants 1) with significant positive changes between the baseline and first post-test measurements, 2) without significant changes, and 3) with negative changes, will be invited for interviews. They will be asked to comment on their experiences and feelings about the intervention that they received and on changes in their behavior, their perceptions of the intervention, their beliefs, concerns, and views of the difficulties of managing pain; and how the intervention could be improved to meet their needs.

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Metropolitan University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No